CLINICAL TRIAL: NCT06805240
Title: EvaluatIng Normal Values for traditionaL anorectaL fUnction paraMeters With aIr Charged aNd Solid State HRAM catheTErs ("ILLUMINATE" Study)
Acronym: ILLUMINATE
Status: Recruiting | Type: Observational
Sponsor: Laborie Medical Technologies Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: CLN-00043; Solar-01 (Other: Laborie Medical Technologies Corporation)
Record Dates: First submitted 2025-01-24; First posted 2025-02-03 (Actual); Last update posted 2025-03-20 (Actual); Status verified 2025-03

CONDITIONS: Healthy
Keywords: ARM procedure; ARM measurement; asymptomatic; Healthy; anorectal function; anorectal

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

INTERVENTIONS:
Diagnostic Test: Air Charged Catheter ARM Procedure — Normative datasets for traditional measures of anorectal function with an air charged HRAM catheter will be collected in healthy subjects using the IAPWG standardized testing protocol and London classification for ARM measurement.
Diagnostic Test: Solid State Catheter ARM Procedure — Normative datasets for traditional measures of anorectal function with a solid state HRAM catheter will be collected in some healthy subjects using the IAPWG standardized testing protocol and London classification for ARM measurement for comparison to the air charged catheter.

SUMMARY:
The research study will be conducted to obtain baseline, or "normative" information to compare an air charged HRAM catheter to traditional solid catheter measures using the IAPWG standardized testing protocol and London classification.

DETAILED DESCRIPTION:
The primary purpose of this research study is to obtain normative datasets for traditional measures of anorectal function with an air charged HRAM catheter in healthy subjects using the IAPWG standardized testing protocol and London classification for anorectal manometry (ARM) measurement.

A secondary purpose is to qualitatively compare the performance of air charged and solid state HRAM catheters in determining values for traditional measures of anorectal function in a subset of study subjects using the IAPWG standardized testing protocol and London classification for ARM measurement.

ELIGIBILITY:
Inclusion Criteria:

* 1. Male and female volunteers, 18-65 years old
* 2. Willing to provide informed consent
* 3. Willing and able to follow instructions for ARM procedure

Exclusion Criteria:

* 1. Documented history of gastrointestinal disorders such as:
* a. fecal incontinence,
* b. irritable bowel syndrome (IBS),
* c. functional constipation, as defined by two or more of these symptoms for at least 25% of the time over the past 3 months:
* i. excessive straining,
* ii. hard or lumpy stools,
* iii. sensation of incomplete evacuation,
* iv. a feeling of anorectal blockage,
* v. manual maneuvers to facilitate defecation,
* vi. or fewer than 3 bowel movements per week.
* d. functional diarrhea, as defined by the following symptoms over the past 3 months:
* i. Loose or watery stools
* ii. Lack of pain with diarrhea
* iii. Diarrhea occurring in at least 75% of bowel movements
* iv. No identifiable causes
* 2. Use of medications that may affect gastrointestinal motility as determined by healthcare professional.
* 3. Prior pelvic radiation,
* 4. Prior anorectal surgical procedures, including treatment for hemorrhoids,
* 5. Risk factors for pelvic floor trauma:
* a. more than 4 vaginal deliveries,
* b. vaginal delivery with birthweight greater than 4500gms (macrosomia),
* c. known 4th degree perineal tear or known forceps use during delivery.
* 6. Contraindicated for ARM testing
* 7. Has gastrointestinal symptoms and is indicated for ARM testing
* 8. Subject is currently pregnant or plans to become pregnant during the course of their enrollment in the study, as self-reported.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy male and female adults, 18-65 years old
Sampling Method: Non-Probability Sample
Enrollment: 81 (Estimated)
Dates: Start 2025-01-09 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Obtain normative datasets | From Baseline to Day 1
  Obtain normative datasets for traditional measures of anorectal function with an air charged HRAM catheter in healthy subjects using the IAPWG standardized testing protocol and London classification for ARM measurement.

SECONDARY OUTCOMES:
Qualitatively compare the performance | From Baseline to Day 1
  Qualitatively compare the performance of air charged and solid state HRAM catheters in determining values for traditional measures of anorectal function in a subset of study subjects using the IAPWG standardized testing protocol and London classification for ARM measurement.

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Augusta University Digestive Health Center, Augusta, Georgia
  - Southwest Gastroenterology, New Lenox, Illinois
  - Digestive Health Center of the Four States, LLC, Joplin, Missouri